CLINICAL TRIAL: NCT02468336
Title: Vascular Reactivity Assessment by a Novel Diagnostic Device, ANGIODEFENDER, Compared to Using Brachial Artery Ultrasound Imaging
Brief Title: AngioDefender Versus Brachial Artery Ultrasound Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Everist Genomics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: A-1302
Record Dates: First submitted 2015-06-07; First posted 2015-06-10 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Cardiovascular Diseases
Keywords: Physiology
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AngioDefender (Experimental): The AngioDefender device uses a novel, proprietary software algorithm to analyze pulse wave amplitude data collected before and after BA occlusion by a standard upper arm sphygmomanometric blood pressure (BP) cuff. The procedure is non-invasive and employs neither ultrasound nor Doppler flow analysis.
  Interventions: Device: AngioDefender
- Brachial Artery Ultrasound Imaging (Active Comparator): A non-invasive procedure for detecting endothelial dysfunction by measuring the flow-mediated dilation of the brachial artery (BA) using high resolution continuous ECG-gated B-mode (2D) ultrasound imaging during reactive hyperemia, a state of transient increase in tissue blood flow that occurs following a brief period of ischemia, e.g., BA occlusion. BA diameter is measured at end-diastole, coincident with the R wave of a simultaneously recorded ECG.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: AngioDefender
  Arms: AngioDefender
Device: Ultrasound
  Arms: Brachial Artery Ultrasound Imaging

SUMMARY:
The objective of this study is to demonstrate that the investigational device, AngioDefender, is comparable to the established procedure referred to as 'brachial artery ultrasound imaging' in their abilities to quantify flow-mediated vasodilation of the brachial artery.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-2

Exclusion Criteria:

1. Body mass index (BMI) >50 kg/m2
2. Mid-upper arm circumference of arm selected for FMD testing <17 cm or >40 cm
3. Sinus arrhythmia (RR intervals vary by >50%), atrial fibrillation, atrial flutter, multifocal atrial tachycardia, frequent (>1 per 10-sec strip) premature atrial or ventricular contractions (isolated, non-isolated, or alternating), documented by 12-lead ECG with rhythm strip at the time of subject screening.
4. Clinical signs and/or symptoms of active viral or bacterial infections
5. Resting tremor or inability to remain still for the duration of AD and BAUI testing
6. Systolic blood pressure (SBP) at rest of >170 mmHg or diastolic blood pressure (DBP) at rest of ≥110 mmHg.
7. Previous intolerable adverse reaction(s) to vascular testing using an upper extremity occlusive pneumatic cuff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Statistical equivalence of %FMD determined by AngioDefender vs brachial artery ultrasound imaging (BAUI) | 1 day
  Deming regression analysis and Bland-Altman Plots

SECONDARY OUTCOMES:
Comparison of types and incidences of emergent adverse device effects | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Peter F Lenehan, MD PhD, Study Director — Everist Health
Locations (5):
- United States (4):
  - University of Colorado, Boulder, Boulder, Colorado
  - Yale University Prevention Research Center, Derby, Connecticut
  - Boston University, Boston, Massachusetts
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No